CLINICAL TRIAL: NCT06127238
Title: A Phase Ib/II Study of ST-1898 to Evaluate the Efficacy and Safety in Patients With Renal Cell Carcinoma (RCC)
Brief Title: Study of ST-1898 in Advanced Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Scitech-Mq Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-1898-201
Record Dates: First submitted 2023-10-22; First posted 2023-11-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: ST-1898, renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 3-(3'-adamantan-1-yl-4'-methoxybiphenyl-4-yl)-2-propenoic acid

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Escalation followed by Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ST-1898 Phase Ib (Experimental): Dose Escalation:participants will be administered orally at 100mg,140mg,160mg,180mg, 220mg,QD during the study, until disease progression or intolerable toxicity.
  Interventions: Drug: ST-1898 tablets
- ST-1898 Phase II (Experimental): Dose Expansion: participants with advanced renal cell carcinoma will be dministered orally at recommended phase II dose from phase Ib once daily during the study, until disease progression or intolerable toxicity.
  Interventions: Drug: ST-1898 tablets

INTERVENTIONS:
Drug: ST-1898 tablets — Supplied as 5 mg and 40 mg tablets

SUMMARY:
ST-1898 is a receptor tyrosine kinase (RTK) inhibitor for multi-targets, especially for VEGFR2, c-MET, AXL，PDGFRA，RET，KIT etc. This trial is to evaluate its safety, tolerability, pharmacokinetic, and efficacy in patients with advanced renal cell carcinoma (RCC).

In phase Ib, the primary objectives are to assess the safety and tolerability, and to determine the maximum tolerated dose (MTD) of ST-1898 tablets in patients with advanced RCC. Secondary objectives are to assess the plasma concentration of ST-1898 and to evaluate the efficacy in patients with advanced RCC.

In phase II, the primary objective is to assess the anti-tumor activities of ST-1898 tablets in patients with advanced RCC. The secondary objective is to evaluate the safety of ST-1898 tablets in patients with advanced RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Life expectancy of three months or more
3. Histologically and medical imaging confirmed unresectable, locally advanced or metastatic renal cell carcinoma. In Dose Escalation Phase, subjects should be progressed with standard therapy, not eligible for standard therapy or no standard therapy available；in Dose Expansion Phase, subjects should be progressed with prior immune checkpoint inhibitor and tyrosine kinase inhibitor therapy.
4. With agreement to provide a tumor tissue specimen
5. Has the ability to understand and willingness to sign a written ICF before the performance of any study-specific procedures on this protocol
6. Has at least one measurable lesion as defined by RECIST version 1.1
7. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
8. Has adequate organ function defined as follows:

   1. Bone marrow : absolute neutrophil count(ANC)≥1.5×10^9 /L, Hb level ≥ 90 g/L and platelet count (PLT) ≥ 90 x10^9/L, no transfusions and no use of colony stimulating factor within 2 weeks prior to routine blood test) at screening;
   2. Liver: transaminase levels (AST/ALT) ≤ 3.0×upper limit of normal (ULN), AST/ALT ≤ 5×ULN for liver metastasis; total bilirubin (TBILI) ≤ 1.5 ×ULN;
   3. Kidney: Creatinine ≤1.5×ULN
   4. Heart: LVEF≥50%
   5. Coagulation function: INR≤1.5×ULN，APTT≤1.5×ULN (except for the prophylactic use of anticoagulants)
   6. Urine protein ≤1+; or in the condition of urine protein ≥2+, quantitative measurement of the 24-hour urine protein is < 1g
9. Women of child bearing potential must have a negative serum pregnancy test within 7 days before first study drug administration. Female patients of child bearing potential, or a male patients with a female partner of child-bearing potential (defined as all women physiologically capable of becoming pregnant), must agree to use a highly effective method of contraception during screening, during the period of drug administration and for 120 days after stopping study drug administration.

Exclusion Criteria:

1. Has received another anti-tumor therapy within two weeks or within 5 half-life of anti- tumor drug prior to the first dose
2. Has had major surgery within 4 weeks before the first study drug administration (except tumor biopsy, puncture, invasive dental procedures such as tooth extraction, dental implants etc.)
3. Current or previous severe retinopathy who, in the judgment of the Investigator or specialist, are not suitable for enrollment
4. Has had any history of major cardiovascular event within 6 months prior to study drug administration including but not limited to :

   1. Serious arrhythmia or cardiac conduct abnormality , such as degree II-III atrioventricular block or ventricular arrhythmia needs to be treated
   2. QTc interval extension: male >450 ms, female >470 ms
   3. Acute coronary syndrome, stroke, deep vein thrombosis, pulmonary- thromboembolism, arterial thrombosis, congestive heart failure, aortic dissection etc.
   4. New York Heart Association Class ≥ II
   5. Has uncontrolled hypertension, as defined by a sustained blood pressure (BP) > 140/90 mmHg with antihypertensive treatment
5. Has brain metastases with symptoms or with evidence of progression
6. Has Interstitial lung disease or radiation pneumonia requiring treatment by steroid
7. Has other malignant tumors in the last 5 years (not including non-melanoma skin cancer, breast cancer or cervical cancer in situ, and Non-Muscle-invasive bladder cancer that have been cured)
8. Has ≥ grade 3 hemorrhage/bleeding event within 6 months prior to study drug administration or currently ≥ grade 2 hemorrhage or event of high risk of hemorrhage) including active gastrointestinal ulcer or esophageal varices
9. Concomitant medication with strong inducers of CYP3A4, strong inhibitors of CYP3A4, or CYP3A4 substrates with narrow therapeutic windows within 2 weeks prior to first dose.
10. Has not recovered from toxicities caused by prior therapy to CTCAE≤ Grade 1 (except for peripheral neuropathy becoming ≤Grade 2, alopecia, and other events judged tolerable by the Investigator and without safety risks).
11. Active hepatitis B (asymptomatic hepatitis B carriers with HBV DNA < 2000 IU/mL are allowed to be enrolled), hepatitis C virus (HCV) antibody-positive and HCV-RNA- positive, or other active hepatitis, clinically significant moderate-to-severe cirrhosis, are allowed to receive prophylactic antiviral therapy other than interferon.
12. Has acute bacterial, viral or fungal infections, requiring systemic anti-infective treatment.
13. HIV positive
14. Pregnant or lactating females
15. Drug or alcohol dependents
16. Has significant disorder of neurology or mental disease or poorly compliance
17. Unable to swallow oral medications or condition or conditions that in the judgment of the Investigator which severely interfere with gastrointestinal absorption, such as dysphagia, intestinal obstruction, etc.
18. Clinically uncontrollable third interstitial effusion that, in the judgment of the Investigator, is unsuitable for enrollment.
19. Has a history of other serious systemic disease, or any other reason that might interfere with participation in trial or interfere with interpretation of trial results, in the judgement of the Investigator, that are not qualified to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib Dose Escalation：Maximum Tolerated Dose (MTD) | Within the first cycle (21days)
  The MTD was defined as the highest dose level at which no more than 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first cycle (21days) of treatment.
Phase Ib Dose Escalation: The Number and frequency of treatment-related adverse events (AEs) and treatment-related serious adverse events (SAEs) | Approximately 18 months
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
Phase II Expansion: Objective Response Rate (ORR) | Approximately 18 months
  ORR is defined as The percentage of participants who experience a CR or PR based on RECIST 1.1 (CR: Complete Response, Disappearance of all target lesions, PR: Partial Response, At least a 30% decrease in the sum of diameters of target lesions)

SECONDARY OUTCOMES:
Phase Ib Dose Escalation: Plasma PK | On Day 1, 8, 21 of Cycle 1 and Day 1 of Cycle 3, approximately 10 weeks
  To assess plasma pharmacokinetics (PK) of oral administration of ST-1898 in participants with advanced renal cell carcinoma
Phase Ib Dose Escalation: ORR | Approximately 18 months
  Objective Response Rate (ORR) per RECIST 1.1
Phase Ib Dose Escalation: DOR | Approximately 18 months
  DOR Duration of Response (DOR) per RECIST 1.1
Phase Ib Dose Escalation: PFS | Approximately 18 months
  Progression-Free Survival (PFS) per RECIST 1.1
Phase Ib Dose Escalation: DCR | Approximately 18 months
  Disease Control Rate (DCR) per RECIST 1.1
Phase Ib Dose Escalation: OS | Approximately 30 months
  Overall Survival (OS)
Phase Ib Dose Escalation: TTP | Approximately 18 months
  Time to Progression（TTP）per RECIST 1.1
Phase II Dose Expansion: DOR | Approximately 18 months
  DOR Duration of Response (DOR) per RECIST 1.1
Phase II Dose Expansion: PFS | Approximately 18 months
  Progression-Free Survival (PFS) per RECIST 1.1
Phase II Dose Expansion: DCR | Approximately 18 months
  Disease Control Rate (DCR) per RECIST 1.1
Phase II Dose Expansion: OS | Approximately 30 months
  Overall Survival (OS) per RECIST 1.1
Phase II Dose Expansion: OS12m | 12 months
  12-Month survival rate（OS12m）
Phase II Dose Expansion: The Number and frequency of treatment-related adverse events and serious adverse events (SAEs) | Approximately 18 months
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Ph D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No